CLINICAL TRIAL: NCT02629926
Title: A Phase IV, Single-Centre, Non-Randomised, Controlled, Open-Label Study to Assess the Use of Growth Hormone (GH) Replacement Therapy (NutropinAq®) During Transition in GH Deficient Survivors of Childhood Cancer to Optimise Somatic Growth & Well-Being
Brief Title: Transitional Growth Hormone (GH) Use in Growth Hormone Deficient (GHD) Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ED07/8440
Record Dates: First submitted 2015-02-09; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Metabolic Diseases; Cancer
MeSH Terms: conditions — Metabolic Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients to receive GH replacement: 30 patients will be recruited to the study who wishes to continue receiving growth hormone replacement, all of whom will receive NutorpinAq Recombinant growth hormone
  Interventions: Other: GH Replacement (NutropinAq®)
- Patients who will not receive GH replacement: An additional 30 patients who elect not to receive growth hormone replacement will provide a parallel control data.
  Interventions: Other: No additional treatment

INTERVENTIONS:
Other: GH Replacement (NutropinAq®) — GH Replacement continued.
  Groups: Patients to receive GH replacement
Other: No additional treatment — GH Replacement not continued.
  Groups: Patients who will not receive GH replacement

SUMMARY:
Cure rates for childhood malignancies have improved at a remarkable pace.With the increasing cure rate came recognition of the long-term detrimental effects of radiotherapy and chemotherapy, known as "late-effects". Endocrine late-effects are particularly prevalent in childhood cancer survivors. Growth Hormone (GH) deficiency is common following radiation to the head and leads to impaired growth, hence GH replacement is given to achieve optimise final height in childhood. In the adult GH is important to maintenance of bone, muscle & fat mass; vascular risk factors; and quality of life. This observational study aims to determine the long-term effect of low dose GH replacement on development of bone, muscle and fat mass; vascular risk; and quality of life in the early years after achievement of final height, a time known as "transition". GH is thought to be essential to development of bone, muscle, and fat mass during this time period.

Patients will be identified in the late -effects endocrine clinic, aged 16-22yrs, who are severely GH deficient. 30 patients will be recruited to the study who wish to continue receiving GH replacement, all of whom will receive recombinant GH. An additional 30 patients who do not wish to receive GH replacement will provide a parallel control data.

All patients will undergo baseline assessment including examination; routine blood tests; urine dipstick; measures on height, weight, waist, and 24 hour blood pressure. Measures will be repeated at six months, and then annually until 25 years of age. Bone density will be measured at baseline, after two years and at age 25yrs. Patients requesting GH replacement will require initial additional visits to teach self injection, then 2-4wkly to assess when correct dose of GH is achieved. The study will enable assessment of the beneficial effects of GH replacement during transition in GH deficient survivors of cancer to be realised.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16--22 years inclusive.
* Both genders.
* Able to provide informed consent.
* Severe GH deficiency (peak GH<5mcg/l on stimulation).
* No GH replacement therapy during the three months preceding the baseline visit.
* Stable anterior pituitary hormone (i.e. sex steroids, hydrocortisone, thyroxine) therapy over the previous six months.
* Life expectancy >24 months.

Exclusion Criteria:

* Acute critical illness (Patients suffering complications following open heart surgery, abdominal surgery, multiple accidental trauma, acute respiratory failure, or similar conditions).
* Active malignant disease (i.e. undergoing active treatment or palliation).
* Patients treated for an intracranial malignancy should have completed therapy two years prior to entering the study.
* Active Cushing's disese or acromegaly
* Pregnancy or desire to conceive within the following year. Patients at risk of pregnancy will be screened by urine pregnancy (HCG) test at the baseline evaluation & treatment initiation visit.
* Breast feeding.
* Proliferative diabetic retinopathy.
* Sensitivity to GH or its preservative

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be identified in the late effects endocrine clinic aged between 16-22 years, which are severely growth hormone deficient.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compare the change in quality of life (QoL) at twelve months with that at baseline for the two treatment groups. For the primary endpoint this will be determined using the GH -specific instrument, the Adult Growth | 12 monthly intervals until the age of 25yrs

SECONDARY OUTCOMES:
compare the change in QoL at each assessment timepoint versus to Baseline for the two treatment groups | 12 monthly intervals until the age of 25yrs
  three generic selfrating questionnaires
Psychological General WellBeing Schedule (PGWBS) | 12 monthly intervals until the age of 25yrs
  Questionnaire completed at 12 months
Shortform 36 (SF36) questionnaire | 12 monthly intervals until the age of 25yrs
  Questionnaire completed at 12 months
EuroQoL 5D (EQ5D) questionnaire | 12 monthly intervals until the age of 25yrs
  AGHDA SF36 PGWBS EQ5D
compare the change in body composition between the two treatment groups at each assessment timepoint versus Baseline. | 12 monthly intervals until the age of 25yrs
  Weight Height Waist & hip circumference Skin thickness Bioimpedance Total body DXA scan
compare the change in cardiovascular risk factors between the two treatment groups at each assessment every 12 months versus Baseline. | 12 monthly intervals until the age of 25yrs
compare the change in bone mineral content between the two treatment groups at each assessment every 12 months versus Baseline. | 12 monthly intervals until the age of 25yrs
compare the change in bone turnover between the two treatment groups at each assessment timepoint versus Baseline. | 12 monthly intervals until the age of 25yrs
  Measurements of:
  DXA Scan
  * Total bone mineral content
  * Bone mineral density at hips and lumbar spine Serum Osteocalcin 24-hour urinary excretion of deoxypyridinoline cross-links
To assess the safety of GH treatment (IGF-I, Blood glucose, HbA1C, Blood pressure, Side effect questionnaire, Adverse events, Scheduled or unscheduled laboratory findings, Changes in concomitant medication) | 12 monthly intervals until the age of 25yrs
  IGF-I Blood glucose HbA1C Blood pressure Side effect questionnaire Adverse events Scheduled or unscheduled laboratory findings Changes in concomitant medication

CONTACTS AND LOCATIONS:
Locations (1):
- The Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom